CLINICAL TRIAL: NCT04540913
Title: A Controlled, Randomized, Double-blinded, Between-subject, Multicenter, Prospective Clinical Study to Evaluate Safety and Effectiveness of RHA® 3 Versus Restylane-L® for Lip Augmentation
Brief Title: RHA® 3 Versus Restylane-L® for Lip Augmentation
Status: Completed | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEO-RHA-1806
Record Dates: First submitted 2020-08-28; First posted 2020-09-07 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Lip Augmentation; Lip
Keywords: Dermal Filler; Hyaluronic acid; Lip; Lip Augmentation
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- RHA 3 (Experimental): Injection of RHA 3 into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Optional touch up treatment provided at 4 Weeks, optional retreatment at 36 or 52 Weeks.
  Interventions: Device: RHA 3
- Restylane- L (Active Comparator): Injection of Restylane- L into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Optional touch up treatment provided at 4 Weeks.
  Interventions: Device: Restylane-L

INTERVENTIONS:
Device: RHA 3 — Investigational Product, RHA® 3 is a viscoelastic, sterile, non-pyrogenic, clear, colorless, homogenous, and biodegradable gel implant. It is formulated with sodium hyaluronic acid (NaHA) at a concentration of 23 mg/g obtained from bacterial fermentation using the Streptococcus equi bacterial strained, crosslinked with 1,4 butanediol diglycidyl ether (BDDE) and reconstituted in a physiological buffer (pH 7.3). RHA® 3 also contains 0.3% lidocaine hydrochloride to reduce pain on injection.
  Arms: RHA 3
Device: Restylane-L — Comparator Product, Restylane-L is a gel of hyaluronic acid generated by Streptococcus species of bacteria, chemically crosslinked with BDDE, stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL with 0.3% lidocaine.
  Arms: Restylane- L

SUMMARY:
This is a multicenter, double-blinded, randomized, prospective, controlled clinical study to identify whether RHA® 3 is non-inferior to Restylane-L® for lip augmentation at Week 12 after the last treatment (initial or touch-up).

At screening, the treating investigator (TI) will evaluate the subject's lip fullness using the validated Teoxane Lip Fullness Scale (5-grade) for eligibility of the subject for the study.

At screening, the blinded live evaluator (BLE) will evaluate the subject's lip fullness using the TLFS to confirm eligibility and to establish a pre-treatment score for assessment of effectiveness.

Enrolled subjects will be randomly assigned in a 3:1 ratio to either the RHA® 3 or the Restylane-L® treatment group. Subjects will be blinded to the study treatment. The TI will administer the fillers, and if necessary, subjects will receive a touch-up treatment 4 weeks after the initial treatment to optimize the results. If the touch-up treatment is administered, the subject will be asked to come to the site for an additional visit 4 weeks after the touch-up injection.

The study duration was extended from 36 to 52 weeks once all subjects had already been enrolled. Nearly 60% of the subjects consented to extend the study to 52 weeks before being eligible for repeat treatment. All data are presented up to 52 weeks (as well as 4 more weeks follow-up after retreatment at 36 or 52 weeks).

Subjects will be followed for 36 to 52 weeks after their last treatment (initial treatment or touch-up), at which point, they will be offered re-treatment with RHA® 3, regardless of their original treatment, provided that the TI deems the treatment to be appropriate and the subject agrees. Reasons for not administering the re-treatment will be documented.

The subject will then be followed for an additional 4 weeks before exiting the study. If the subject or the TI declines re-treatment, this visit (36 or 52 weeks after the last treatment) will be considered the study Exit visit.

For subjects with re-treatment, the Exit visit will be 4 weeks after the re-treatment.

The TI will conduct safety and effectiveness evaluations at each study visit (up to 36 weeks or 52 (if applicable) weeks after the last treatment, and 4 weeks after re treatment) or until all treatment-related ongoing adverse events (AEs) have resolved or resolved with sequelae as per TI judgment or if follow-up is no longer possible.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, 22 years of age or older
* Lip fullness of grade 1 to 3 on the TLFS (ranging from 1 to 5) who desire at least 1 point of correction for upper and/or lower lips OR has Fitzpatrick skin type V or VI and has lip fullness grade 4 or 5 on the TLFS who desire treatment to the vermillion body for upper and/or lower lips. The BLE and TI must independently assess and agree that this criterion is met; however, concordance of fullness is not required. If the assessments of the TI and the BLE are the same or differ by exactly 1 point on the scale, this difference is considered acceptable. If the assessments differ by 2 points or more on the scale, the subject will not be eligible.
* Willing to abstain from facial aesthetic procedures/therapies that could interfere with study evaluations
* Able to follow study instructions and complete all required visits.
* Sign the IRB-approved ICF, Photographic Release Form and the Authorization for Use and release of Health and Research Study Information (HIPAA) form prior to any study- related procedures being performed.

Exclusion Criteria:

* Female subjects that are pregnant, breast-feeding or of childbearing potential and not practicing reliable birth control
* Known hypersensitivity/allergy to any component of the study devices
* Clinically significant active skin disease within 6 months
* Has a history of or currently has an auto-immune disease.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- United States, Florida, Bradenton, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- RHA 3: Injection of RHA 3 into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Optional touch up treatment provided at 4 Weeks, optional retreatment at 36 or 52 Weeks.
  RHA 3: Investigational Product, RHA® 3 is a viscoelastic, sterile, non-pyrogenic, clear, colorless, homogenous, and biodegradable gel implant. It is formulated with sodium hyaluronic acid (NaHA) at a concentration of 23 mg/g obtained from bacterial fermentation using the Streptococcus equi bacterial strained, crosslinked with 1,4 butanediol diglycidyl ether (BDDE) and reconstituted in a physiological buffer (pH 7.3). RHA® 3 also contains 0.3% lidocaine hydrochloride to reduce pain on injection.
- Control Device: Injection of control device into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Optional touch up treatment provided at 4 Weeks.
  Comparator Product: a gel of hyaluronic acid generated by Streptococcus species of bacteria, chemically crosslinked with BDDE, stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL with 0.3% lidocaine.
Period: Overall Study
Arm/Group | RHA 3 | Control Device
Started | 153 | 49
ITT Population | 148 | 48
mITT Population | 137 | 44
PP Population | 127 | 42
Completed | 139 | 46
Not Completed | 14 | 3
Not completed — Withdrawal by Subject | 14 | 3

BASELINE CHARACTERISTICS:
Groups:
- RHA 3: Injection of RHA 3 into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Optional touch up treatment provided at 4 Weeks, retreatment at 36 or 52 Weeks.
  RHA 3: Investigational Product, RHA® 3 is a viscoelastic, sterile, non-pyrogenic, clear, colorless, homogenous, and biodegradable gel implant. It is formulated with sodium hyaluronic acid (NaHA) at a concentration of 23 mg/g obtained from bacterial fermentation using the Streptococcus equi bacterial strained, crosslinked with 1,4 butanediol diglycidyl ether (BDDE) and reconstituted in a physiological buffer (pH 7.3). RHA® 3 also contains 0.3% lidocaine hydrochloride to reduce pain on injection.
- Restylane- L: Injection of Restylane- L into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Optional touch up treatment provided at 4 Weeks.
  Restylane-L: Comparator Product, Restylane-L is a gel of hyaluronic acid generated by Streptococcus species of bacteria, chemically crosslinked with BDDE, stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL with 0.3% lidocaine.
- Total: Total of all reporting groups
Arm/Group | RHA 3 | Restylane- L | Total
Number analyzed (Participants) | 153 | 49 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (13.19) | 48.5 (11.69) | 48.7 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 48 | 199
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 15 | 2 | 17
  White | 130 | 45 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 153 | 49 | 202
Fitzpatrick Skin Type [1] [Count of Participants; unit: Participants] — Fitzpatrick skin type as determined by the Treating Investigator on the skin tone scale developed to classify skin coloring and response to ultraviolet (UV) radiation. The scale contains 6 grades:
  I: Pale white skin; Always burns, does not tan. II: Fair skin; Burns easily, tans poorly. III: Darker white skin; Tans after initial burn. IV: Light brown skin; Burns minimally, tans easily. V: Brown skin; Rarely burns, tans darkly easily. VI: Dark brown or black skin; Never burns, always tans darkly.
  Participants
    Type I-III | 114 | 35 | 149
    Type IV-VI | 39 | 14 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in TLFS Score (Teoxane Lip Fullness Scale) Between Baseline and Week 12 After Last Treatment of RHA®3 Versus Control Device, as Assessed by the BLE
Description: A change in the TLFS ≥1 grade compared to pre-treatment will be considered clinically meaningful.
  The TLFS is a validated 5-point scale for assessing lip augmentation. Possible scores range from 1 (Very Thin) to 5 (Very Full).
  Change = (Week 12 - Baseline score).
Time Frame: Week 12 after last treatment
Population: Primary endpoint on the mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Device: Injection of control device into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Optional touch up treatment provided at 4 Weeks.
  Control Device: a gel of hyaluronic acid generated by Streptococcus species of bacteria, chemically crosslinked with BDDE, stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL with 0.3% lidocaine.
Arm/Group | RHA 3 | Control Device
Number analyzed (Participants) | 137 | 44
score on a scale | 1.0 (0.65) | 0.8 (0.70)

2. Secondary Outcome: Change From Baseline in TLFS Score as Assessed by the BLE at Visit 5 (Weeks 24 After Last Treatment), 6 (Weeks 36 After Last Treatment), 7 (Week 52 After Last Treatment) if Applicable, and Re-treatment (4 Weeks After Re-treatment)
Description: A change in the TLFS ≥1 grade compared to pre-treatment will be considered clinically meaningful.
  The TLFS is a validated 5-point static scale for assessing lip augmentation. Possible scores range from 1 (Very Thin) to 5 (Very Full).
Time Frame: Weeks 36 and 52 after last treatment, week 4 after re-treatment
Population: mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA 3 | Control Device
Number analyzed (Participants) | 137 | 44
score on a scale
  Week 36 after last treatment: number analyzed (Participants) | 132 | 43
  Week 36 after last treatment | 0.7 (0.65) | 0.5 (0.63)
  Week 52 after last treatment: number analyzed (Participants) | 79 | 23
  Week 52 after last treatment | 0.5 (0.64) | 0.1 (0.63)
  Re-treatment: 4weeks post re-treatment at week 36: number analyzed (Participants) | 23 | 10
  Re-treatment: 4weeks post re-treatment at week 36 | 1.0 (0.82) | 0.9 (0.74)
  Re-treatment: 4 weeks post re-treatment at week 52: number analyzed (Participants) | 59 | 17
  Re-treatment: 4 weeks post re-treatment at week 52 | 1.1 (0.74) | 0.9 (0.66)

3. Secondary Outcome: Responder Rate Calculated Using TLFS Assessed by the BLE
Description: A responder will be defined as a subject who has a ≥1 grade improvement on the TLFS.
  The TLFS is a validated 5-point static scale for assessing lip augmentation. Possible scores range from 1 (Very Thin) to 5 (Very Full).
Time Frame: Weeks 12, 36, 52 after last treatment, week 4 after re-treatment
Population: mITT population
Measure: Count of Participants; unit: Participants
Groups:
- Control Device: Injection of control device into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Optional touch up treatment provided at 4 Weeks.
  Comparator Product is a gel of hyaluronic acid generated by Streptococcus species of bacteria, chemically crosslinked with BDDE, stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL with 0.3% lidocaine.
Arm/Group | RHA 3 | Control Device
Number analyzed (Participants) | 137 | 44
Participants
  Week 12 after last treatment: number analyzed (Participants) | 135 | 43
  Week 12 after last treatment | 105 | 29
  Week 36 after last treatment: number analyzed (Participants) | 132 | 43
  Week 36 after last treatment | 81 | 22
  Week 52 after last treatment: number analyzed (Participants) | 79 | 23
  Week 52 after last treatment | 38 | 6
  Re-treatment: 4weeks post re-treatment at week 36: number analyzed (Participants) | 23 | 10
  Re-treatment: 4weeks post re-treatment at week 36 | 18 | 7
  Re-treatment: 4weeks post re-treatment at week 52: number analyzed (Participants) | 59 | 17
  Re-treatment: 4weeks post re-treatment at week 52 | 49 | 13

4. Secondary Outcome: Number of Subjects "Satisfied" or "Very Satisfied" With Study Treatment Using the Subject Satisfaction Scale at Weeks 12, 36, 52 After Last Treatment and 4 Weeks After Re-treatment.
Description: The Subject Satisfaction Scale is a subjective, balanced, 5-point scale assessing subject satisfaction with study treatment. Possible scores range from with 1 (very satisfied) to 5 (very dissatisfied).
Time Frame: Weeks 12, 36, 52 after last treatment and 4 week after re-treatment.
Population: mITT population
Measure: Count of Participants; unit: Participants
Groups:
- Restylane-L: Injection of control device into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Optional touch up treatment provided at 4 Weeks.
  Comparator Product is a gel of hyaluronic acid generated by Streptococcus species of bacteria, chemically crosslinked with BDDE, stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL with 0.3% lidocaine.
Arm/Group | RHA 3 | Restylane-L
Number analyzed (Participants) | 137 | 44
Participants
  Week 12 after last treatment: number analyzed (Participants) | 135 | 43
  Week 12 after last treatment | 113 | 33
  Week 36 after last treatment: number analyzed (Participants) | 132 | 43
  Week 36 after last treatment | 108 | 27
  Week 52 after last treatment: number analyzed (Participants) | 81 | 23
  Week 52 after last treatment | 67 | 16
  Re-treatment: 4 weeks post re-treatment at week 36: number analyzed (Participants) | 23 | 10
  Re-treatment: 4 weeks post re-treatment at week 36 | 22 | 9
  Re-treatment: 4 weeks post re-treatment at week 52: number analyzed (Participants) | 59 | 17
  Re-treatment: 4 weeks post re-treatment at week 52 | 54 | 15

5. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the "Satisfaction With Lips" FACE-Q | Aesthetics© Scale Questionnaire at Weeks 12, 36, 52 After Last Treatment and 4 Week After Re-treatment.
Description: The FACE-Q measures the experience and outcomes of aesthetic facial procedures from the patient's perspective.
  The FACE-Q questionnaire is composed of 10 questions with a score linked to answers (1 being "Very Dissatisfied" and 4 being "Very Satisfied").
  The subject will be instructed as follows: "These questions ask about how you look right now. For each question, circle only one answer. With your lips in mind, in the past week, how satisfied or dissatisfied have been with:", and will provide response.
  To calculate the FACE-Q, outcomes from all 10 questions were pooled, data were transformed so that higher scores reflected a superior (positive) outcome, and adapted to a scale of 100 units (i.e. worst/lowest score = 0, best/highest score = 100).
Time Frame: Change from Baseline at Weeks 12, 36, 52 after last treatment and 4 week after re-treatment.
Population: mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA 3 | Restylane-L
Number analyzed (Participants) | 137 | 44
score on a scale
  Week 12 after last treatment: number analyzed (Participants) | 135 | 43
  Week 12 after last treatment | 50.6 (25.58) | 46.1 (26.71)
  Week 36 after last treatment: number analyzed (Participants) | 132 | 43
  Week 36 after last treatment | 40.9 (29.11) | 31.8 (30.76)
  Week 52 after last treatment: number analyzed (Participants) | 81 | 23
  Week 52 after last treatment | 36.2 (27.56) | 25.1 (30.60)
  Re-treatment: 4weeks post re-treatment at week 36: number analyzed (Participants) | 23 | 10
  Re-treatment: 4weeks post re-treatment at week 36 | 57.4 (24.42) | 55.7 (19.7)
  Re-treatment: 4weeks post re-treatment at week 52: number analyzed (Participants) | 60 | 17
  Re-treatment: 4weeks post re-treatment at week 52 | 56.0 (23.8) | 51.9 (20.45)

6. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the "Satisfaction With Outcome" FACE-Q | Aesthetics© Scale Questionnaire at Weeks 12, 36, 52 After Last Treatment and 4 Week After Re-treatment.
Description: The FACE-Q measures the experience and outcomes of aesthetic facial procedures from the patient's perspective.
  The FACE-Q questionnaire is composed of 6 questions with a score linked to answers (1 being "Definitely disagree" and 4 being "Definitely agree").
  The subject will be instructed as follows: "We would like to know how you feel about your most recent procedure. For each question, select only one answer. Please indicate how much you agree or disagree with each statement:", and will provide response.
  To calculate the FACE-Q, outcomes from all 16questions were pooled, data were transformed so that higher scores reflected a superior (positive) outcome, and adapted to a scale of 100 units (i.e. worst/lowest score = 0, best/highest score = 100).
Time Frame: Weeks 12, 36, 52 after last treatment and 4 week after re-treatment.
Population: mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA 3 | Restylane-L
Number analyzed (Participants) | 137 | 44
score on a scale
  Week 12 after last treatment: number analyzed (Participants) | 135 | 43
  Week 12 after last treatment | 77.2 (22.65) | 71.1 (29.64)
  Week 36 after last treatment: number analyzed (Participants) | 132 | 43
  Week 36 after last treatment | 73.8 (26.03) | 61.9 (33.62)
  Week 52 after last treatment: number analyzed (Participants) | 81 | 23
  Week 52 after last treatment | 75.6 (24.08) | 61.6 (30.65)
  Re-treatment: 4weeks post re-treatment at week 36: number analyzed (Participants) | 23 | 10
  Re-treatment: 4weeks post re-treatment at week 36 | 81.0 (19.43) | 76.8 (22.84)
  Re-treatment: 4weeks post re-treatment at week 52: number analyzed (Participants) | 60 | 17
  Re-treatment: 4weeks post re-treatment at week 52 | 82.4 (20.61) | 75.6 (27.5)

7. Secondary Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the BLE.
Description: The Global Aesthetic Improvement (GAI) is a subjective, balanced, 5-point dynamic scale assessing cosmetic improvement.
  Possible scores range from "much improved", "improved", "no change", "worse", to "much worse". The GAI will be assessed using the baseline photograph.
Time Frame: Weeks 12, 36, 52 after last treatment, and 4 weeks after re-treatment
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | RHA 3 | Control Device
Number analyzed (Participants) | 137 | 44
Participants
  Week 12 after last treatment: number analyzed (Participants) | 135 | 43
  Week 12 after last treatment | 134 | 41
  Week 36 after last treatment: number analyzed (Participants) | 132 | 43
  Week 36 after last treatment | 113 | 29
  Week 52 after last treatment: number analyzed (Participants) | 79 | 23
  Week 52 after last treatment | 58 | 11
  Re-treatment: 4weeks post re-treatment at week 36: number analyzed (Participants) | 23 | 10
  Re-treatment: 4weeks post re-treatment at week 36 | 21 | 8
  Re-treatment: 4weeks post re-treatment at week 52: number analyzed (Participants) | 59 | 17
  Re-treatment: 4weeks post re-treatment at week 52 | 58 | 17

ADVERSE EVENTS:
Time Frame: 36 to 44 (for patients receiving re-treatment) weeks for subjects who did not consent to study extension. 52 to 60 (for patients receiving re-treatment) weeks for subjects who consented to the study extension
Groups:
- RHA 3: Injection of RHA 3 into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Touch up treatment provided at 4 Weeks, retreatment at 36 or 52 Weeks.
  RHA 3: Investigational Product, RHA® 3 is a viscoelastic, sterile, non-pyrogenic, clear, colorless, homogenous, and biodegradable gel implant. It is formulated with sodium hyaluronic acid (NaHA) at a concentration of 23 mg/g obtained from bacterial fermentation using the Streptococcus equi bacterial strained, crosslinked with 1,4 butanediol diglycidyl ether (BDDE) and reconstituted in a physiological buffer (pH 7.3). RHA® 3 also contains 0.3% lidocaine hydrochloride to reduce pain on injection.
- Restylane- L: Injection of Restylane- L into into the vermillion body, vermillion border, and oral commissures of the lips (up to 3 ml with a max of 1.5 ml per lip), injected into the lip mucosa and/or mid to deep dermis as appropriate for lip augmentation.
  Touch up treatment provided at 4 Weeks.
  Restylane-L: Comparator Product, Restylane-L is a gel of hyaluronic acid generated by Streptococcus species of bacteria, chemically crosslinked with BDDE, stabilized and suspended in phosphate buffered saline at pH=7 and concentration of 20 mg/mL with 0.3% lidocaine.
Arm/Group | RHA 3 | Restylane- L
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/153 | 1/49
Other Adverse Events (participants affected / at risk) | 75/153 | 22/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHA 3 (N=153) | Restylane- L (N=49)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.65% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHA 3 (N=153) | Restylane- L (N=49)
Injection Site Mass (General disorders) | 29 (36) | 11 (14)
Injection Site Swelling (General disorders) | 17 (19) | 6 (7)
Injection Site Induration (General disorders) | 14 (18) | 5 (6)
Injection Site Bruising (General disorders) | 8 (8) | 1 (1)
Injection Site Pain (General disorders) | 5 (5) | 4 (4)
Injection Site Erosion (General disorders) | 5 (6) | 3 (4)
Injection Site Reaction (General disorders) | 6 (7) | 2 (2)
Injection Site Deformation (General disorders) | 7 (8) | 0 (0)
Injection Site Exfoliation (General disorders) | 4 (6) | 2 (4)
Injection Site Hypoaesthesia (General disorders) | 4 (8) | 0 (0)
Injection Site Discolouration (General disorders) | 3 (3) | 0 (0)
Injection Site Movement Impairment (General disorders) | 2 (2) | 1 (1)
Injection Site Discomfort (General disorders) | 2 (2) | 0 (0)
Injection Site Dryness (General disorders) | 2 (2) | 0 (0)
Injection Site Hyperaesthesia (General disorders) | 2 (2) | 0 (0)
Injection Site Paraesthesia (General disorders) | 2 (3) | 0 (0)
Injection Site Scab (General disorders) | 1 (1) | 1 (1)
Swelling Face (General disorders) | 0 (0) | 2 (2)
Injection Site Haemorrhage (General disorders) | 0 (0) | 1 (1)
Injection Site Vesicles (General disorders) | 0 (0) | 1 (2)
Covid-19 (Infections and infestations) | 9 (9) | 2 (2)
Injection Site Infection (Infections and infestations) | 3 (5) | 1 (1)
Oral Herpes (Infections and infestations) | 3 (3) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 12 (14) | 5 (5)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial Aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chapped Lips (Gastrointestinal disorders) | 2 (2) | 0 (0)
Salivary Gland Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT04540913/Prot_004.pdf
  • Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT04540913/SAP_005.pdf